CLINICAL TRIAL: NCT07407660
Title: Shortened Venetoclax Duration Based on Bone Marrow Blasts on Day 14 Versus Standard Therapy in Elderly or Frail Patients With Acute Myeloid Leukemia Treated With Azacitidine Plus Venetoclax: A Multicenter Prospective Randomized Controlled Study
Brief Title: Shortened Venetoclax Duration Based on Day 14 BM Blasts Versus Standard Therapy in Elderly or Frail Patients With AML Patients Treated With Azacitidine Plus Venetoclax
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai Qianzhanruiji Enterprise Consulting Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Qian Jiang, Deputy director, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-h243
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Venetoclax; Azacitidine; Early assessment; Treatment optimization; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized treatment (Experimental): Bone marrow aspiration is perfomed on day 14 of the first induction cycle. If the bone marrow blast count is <5%, the duration of venetoclax will be shortened to 14 days; otherwise, the 28-day course will be completed.
  In the second cycle, patients who fail to achieve CR/CRi and those who achieve CR will receive a 28-day course of venetoclax plus azacitidine; for patients who achieve CRi, a 21-day course of venetoclax plus azacitidine will be administered within 14 days following the first cycle.
  Treatment for subsequent cycles will be determined according to the investigators' local clinical practice, including but not limited to continued venetoclax-azacitidine therapy, switching to intensive chemotherapy, or allogeneic hematopoietic stem cell transplantation.
  Interventions: Drug: Venetoclax; Drug: Azacitidine (AZA)
- Standard treatment (Active Comparator): No bone marrow assessment was performed on day 14 of the first induction cycle. All the patients receive the 28-day course of venetoclax plus azacitidine for the first cycle.
  In the second cycle, patients who fail to achieve CR/CRi and those who achieve CR will receive a 28-day course of venetoclax plus azacitidine; for patients who achieve CRi, a 21-day course of venetoclax plus azacitidine will be administered within 14 days following the first cycle.
  Treatment for subsequent cycles will be determined according to the investigators' local clinical practice, including but not limited to continued venetoclax-azacitidine therapy, switching to intensive chemotherapy, or allogeneic hematopoietic stem cell transplantation.
  Interventions: Drug: Venetoclax; Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: Venetoclax — Tablet
Drug: Azacitidine (AZA) — Solution for subcutaneous

SUMMARY:
This study aims to compare the efficacy and safety of a shortened treatment course based on the bone marrow blast count on Day 14 versus standard treatment in patients with acute myeloid leukemia treated with venetoclax plus azacitidine.

DETAILED DESCRIPTION:
The standard 28-day cycle of venetoclax is widely recommended for the first cycle of venetoclax plus azacitidine induction therapy in patients with acute myeloid leukemia (AML). However, it has been found that the 28-day treatment cycle was not tolerant for some patients due to severe myelosuppression and infection, which may lead to treatment interruption and delays in subsequent treatment cycles.

This is a multicenter, randomized controlled, open-label, non-inferiority study, which compare the efficacy and safety of a shortened treatment course based on the bone marrow blast count on Day 14 versus standard treatment in AML patients treated with venetoclax plus azacitidine induction therapy.

This study plans to enroll 250 newly diagnosed AML patients who are intolerant to intensive chemotherapy regimens. Enrolled subjects will be assigned to either the optimized treatment group or the standard treatment group in a 1:1 ratio with stratified blocked randomization, with ELN 2022 classification as the stratification factor. In the optimized treatment group, if the bone marrow blast count is <5% on Day 14 of the first induction, the duration of venetoclax will be shortened to 14 days; otherwise, the 28-day course will be completed as scheduled. In the standard treatment group, no bone marrow assessment will be performed on Day 14, and all patients will complete the 28-day treatment course. The duration of venetoclax in the second cycle will be 28 days or 21 days (if complete remission with incomplete hematologic recovery) for the two groups. The primary endpoint is the achievement of complete remission or complete remission with incomplete hematologic recovery (CR/CRi) within 2 treatment courses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed acute myeloid leukemia who meet the WHO 2022 criteria.
2. Meeting one of the following conditions:

   1. Aged ≥ 60 years;
   2. aged ≥ 18 years and < 60 years, with one or more of the following comorbidities that render the subject unsuitable for intensive induction therapy:

      * Complicated with congestive heart failure, or left ventricular ejection fraction ≤ 50%, or a history of chronic stable angina pectoris;
      * A history of pulmonary disease, with carbon monoxide diffusing capacity of the lung (DLCO) ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%;
      * Creatinine clearance rate < 45 mL/min (calculated by the **Cockcroft-Gault formula**);
      * Total bilirubin > 1.5 × upper limit of normal;
      * Eastern Cooperative Oncology Group (ECOG) performance status (PS) score ≥ 2;
      * Any other comorbidities judged by the investigator to contraindicate intensive induction therapy.
3. Received induction therapy with the azacitidine plus venetoclax regimen (azacitidine for injection: 75 mg/m² subcutaneously on Days 1-7; venetoclax tablets: 100 mg on Day 1, 200 mg on Day 2, and 400 mg once daily starting on Day 3) for 12-14 days. Dose adjustment of venetoclax shall be performed if combined with strong or moderate CYP3A/P-gp inhibitors.
4. Completed risk stratification assessment per the ELN 2022 criteria.
5. Signed the informed consent form.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia, AML with t(8;21)(q22;q22.1)/ RUNX1::RUNX1T1 translocation, or blast crisis of chronic myeloid leukemia (CML).
2. Prior treatment with venetoclax before the diagnosis of acute myeloid leukemia.
3. A history of allogeneic hematopoietic stem cell transplantation.
4. Severe hepatic or renal impairment, defined by the presence of any of the following abnormalities: aspartate aminotransferase (AST) > 2.5 × ULN; alanine aminotransferase (ALT) > 2.5 × ULN; creatinine clearance rate < 30 mL/min (calculated by the Cockcroft-Gault formula); or total bilirubin > 3 × ULN.
5. Presence of acute active infection requiring intravenous systemic therapy.
6. Presence of active malignant tumors requiring antineoplastic treatment.
7. Presence of active autoimmune diseases requiring treatment with prednisone ≥ 15 mg/day or equivalent doses of other glucocorticoids, or any other immunosuppressive agents.
8. Inability to swallow tablets, or presence of diseases significantly impairing gastrointestinal function (e.g., malabsorption syndrome, gastrectomy or enterectomy, bariatric surgery, symptomatic inflammatory bowel disease, or partial/complete intestinal obstruction).
9. Pregnant or lactating female subjects.
10. Subjects judged by the investigator to be unable to comply with the protocol due to uncontrollable medical, psychological, familial, social, or geographic conditions; or those who are unwilling or unable to follow the required procedures of the protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of CR/CRi within 2 treatment cycles | At the end of Cycle 1 and Cycle 2 (each cycle is 28 days). If CRi, repeat 2 weeks later.

SECONDARY OUTCOMES:
Achievement of CR within 2 treatment cycles | At the end of Cycle 1 and Cycle 2 (each cycle is 28 days). If CRi, repeat 2 weeks later.
Achievement of CR/CRi during treatment with the venetoclax plus azacitidine regimen | At the end of Cycles 1, 2, 3, and 5 (each cycle is 28 days) of the venetoclax-azacitidine regimen, and every 2 cycles thereafter.
Achievement of MRD negativity during treatment with the venetoclax plus azacitidine regimen | At the end of Cycles 1, 2, 3, and 5 (each cycle is 28 days) of the venetoclax-azacitidine regimen, and every 2 cycles thereafter.
  Flow cytometry analysis of bone marrow specimen.
Relapse-free survival | From the first achievement of CR/CRi to disease relapse or death from any cause, whichever came first, assessed up to 48 months.
  Relapse-free survival is defined as the number of months from the first achievement of CR/CRi to disease relapse or death from any cause, whichever came first, or censored at the last follow-up.
Overall survival | Time from enrollment to death from any cause, assessed up to 48 months.
  Overall survival is defined as the number of months from enrollment to death from any cause, or censored at the last follow-up.
Adverse events | Time from enrollment to the end of the 2nd treatment cycle (each cycle is 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, Dr., Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF